CLINICAL TRIAL: NCT03612427
Title: Diastolic Blood Pressure and Lipid Profile in Breastfed Vs. Formula Fed Infants ( As Early Indicators for Cardiovascular Disease ).
Brief Title: Diastolic Blood Pressure and Lipid Profile in Infants
Acronym: ERAhmed
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El-Shazly Rabeeh Ahmed, Principal Investigator, Assiut University
Other Study IDs: ERAhmed AssiutU
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Breastfeeding, Exclusive
MeSH Terms: conditions — Breast Feeding | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breastfed infants: Infants depending on breastfeeding S. Cholesterol S. Triglycerides S. HDL Cholesterol
  Interventions: Dietary Supplement: S. Cholesterol S. Triglyceride
- Formula-fed infants: Infants have formula feeding S. Cholesterol S. Triglycerides S. HDL Cholesterol
  Interventions: Dietary Supplement: S. Cholesterol S. Triglyceride

INTERVENTIONS:
Dietary Supplement: S. Cholesterol S. Triglyceride — S. Cholesterol S. Triglycerides
  Other Names: Blood pressure

SUMMARY:
The influence of early environmental factors, including nutrition, on future cardiovascular disease (CVD) risk and, in a broader view, the concept of early metabolic programming and future health have been extensively discussed during the past decades. Observational studies have suggested that formula-fed infants as compared with breastfed infants have an elevated risk of future CVD.

DETAILED DESCRIPTION:
The influence of early environmental factors, including nutrition, on future cardiovascular disease (CVD) risk and, in a broader view, the concept of early metabolic programming and future health have been extensively discussed during the past decades. Observational studies have suggested that formula-fed infants as compared with breastfed infants have an elevated risk of future CVD, since they have faster early growth rate and higher risk of overweight, type 2 diabetes, high blood pressure, and unfavorable blood lipid profile in adult age. Formula-fed preterm infants have higher serum C-reactive protein (CRP) concentration, higher serum low-density lipoprotein to high-density lipoprotein (LDL:HDL) ratio, and higher serum apolipoprotein B to apolipoprotein A1 (apoB:apoA1) ratio in adolescence as compared with preterm infants receiving banked breast milk.

ELIGIBILITY:
Inclusion Criteria:

1. Breastfed infants
2. Formula-fed infants
3. Raw milk fed infants
4. Mixed fed infants

   1. Breast milk plus raw milk
   2. Breast milk plus formula

Exclusion Criteria:

1. Children with Cong. Heart Disease, family history of congenital hyperlipidemia and cases which prove hyperlipidemia of high levels (congenital).

Ages: 10 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients will be recruited outpatient clinic of Assiut pediatric hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Diastolic blood pressure | Around one year
  Value of Infants feeding

SECONDARY OUTCOMES:
Serum cholesterol level | Around one year
  Value of breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: El-Shazly Ahmed, MBBCh, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No